CLINICAL TRIAL: NCT03452982
Title: Sentinel Lymph Node in Early Ovarian Cancer
Acronym: SENTOV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SENTOV
Record Dates: First submitted 2018-02-12; First posted 2018-03-02 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Cancer
Keywords: SENTINEL LYMPH NODE
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Controlled, prospective, descriptive and not randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ovarian cancer (Experimental): Injection of a tracer in the stump of the infundibulo-pelvic ligament and uterus-ovary for sentinel node detection
  Interventions: Other: sentinel node technique

INTERVENTIONS:
Other: sentinel node technique — Injection of a tracer in the stump of the infundibulo-pelvic ligament and uterus-ovary for sentinel node detection.

SUMMARY:
This research study evaluates the concordance of the result between two diagnostic tests: Sentinel node and Pelvic-para-aortic lymphadenectomy in patients with ovarian cancer.

DETAILED DESCRIPTION:
The objective of this study is to describe the feasibility of performing the sentinel node technique (Detection rate) in patients with early stage ovarian cancer.

With this research study it will be evaluated the concordance of the result between two diagnostic tests: Sentinel node and Pelvic-para-aortic lymphadenectomy in patients with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed previously to performing any procedure related to the clinical trial.
* Patients who are women 18 years of age or older at the moment of the randomization.
* Patients with anatomopathological diagnosis of malignant ovarian tumor in a deferred study proposals for staging surgery or patients with suspicious tumor of malignancy who are going to be subjected to exploratory lapaotomy or laparoscopy and operative biopsy, and in the case this is positive, surgery of staging will be performed .

Exclusion Criteria:

* Informed consent not obtained or withdraw.
* Benign result in extemporaneous study
* Previous history of vascular surgery in the aorta, cava or pelvic vessels
* Previous pelvic or para-aortic lymphadenectomy
* Previous lymphoma
* Previous abdomino-pelvic tumor
* Previous allergic reaction to indocyanine green
* Pregnancy / lactation
* Severe adherent syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of performing the sentinel node technique (Detection rate) | Intraoperative (day 0)
  The objective of this study is to describe the feasibility of performing the sentinel node technique (Detection rate) in patients with previous ovarian surgery injecting the tracer in the stump of the infundibulo-pelvic ligament and uterus-ovary for sentinel node detection.

SECONDARY OUTCOMES:
Rate of realization of the technique | Intraoperative (day 0)
Rate of realization of the technique | After anatomopathological study (day 30)
Anatomical location of the sentinel node(s) | Intraoperative (day 0)
  Assessed by radiation (99Tc-nanocoloides) and staining with indocyanine green
Anatomical location of the sentinel node(s) | After anatomopathological study (day 30)
  Assessed by the pathologist
Number of detected sentinel nodes | Intraoperative (day 1)
Number of detected sentinel nodes | After anatomopathological study (day 30)
Characterization of the sample by collecting baseline characteristics | Screening (day 0)
  Age (years)
Characterization of the sample by collecting baseline characteristics | Screening (day 0)
  Weight (kilograms)
Characterization of the sample by collecting baseline characteristics | Screening (day 0)
  Height (centimeters)
Characterization of the sample by collecting baseline characteristics | Screening (day 0)
  BMI (kg/m^2)
Characterization of the sample by collecting baseline characteristics | Screening (day 0)
  Previous gynecological surgery and previous pathological anatomy
Characterization of the sample by collecting tumor markers | Day 0
  Ca 125 and Ca 19.9.
Characterization of the sample by collecting intraoperative findings | Day 0
  Ascites (milliliters)
Characterization of the sample by collecting intraoperative findings | Day 0
  Tumor size (centimeters) of: right ovary, left ovary, right tube, left tube, uterus, pelvic nodes, para-aortic nodes, and tumor in upper hemiabdomen.
Characterization of the sample by collecting surgical procedures | Day 0
  Hysterectomy, adnexectomy, appendectomy, peritonectomy / peritoneal biopsy, omentectomy, lymphadenectomy and blood transfusion (Realized or Unrealized)
Characterization of the sample by collecting surgical procedures | Day 0
  Intraoperative complications
Characterization of the sample by collecting surgical procedures | Day 0
  Result of intraoperative biopsy (unrealized, malignant, benign)
Characterization of the sample by collecting surgical procedures | Day 0
  Estimated blood loss (milliliters)
Characterization of the sample by collecting surgical procedures | Day 0
  Surgical time (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lago, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lago V, Montero B, Lopez S, Padilla-Iserte P, Matute L, Marina T, Gurrea M, Montoliu G, Bello P, Domingo S. Ultrastaging protocol in sentinel lymph node for apparent early stage ovarian cancer. Gynecol Oncol. 2021 May;161(2):408-413. doi: 10.1016/j.ygyno.2021.03.001. Epub 2021 Mar 10. PMID 33712275
- [Derived] Lago V, Bello P, Montero B, Matute L, Padilla-Iserte P, Lopez S, Marina T, Agudelo M, Domingo S. Sentinel lymph node technique in early-stage ovarian cancer (SENTOV): a phase II clinical trial. Int J Gynecol Cancer. 2020 Sep;30(9):1390-1396. doi: 10.1136/ijgc-2020-001289. Epub 2020 May 23. PMID 32448808
- [Derived] Lago V, Bello P, Matute L, Padilla-Iserte P, Marina T, Agudelo M, Domingo S. Sentinel Lymph Node Technique in Apparent Early Ovarian Cancer: Laparoscopic Technique. J Minim Invasive Gynecol. 2020 Jul-Aug;27(5):1019-1020. doi: 10.1016/j.jmig.2019.09.790. Epub 2019 Oct 16. PMID 31628986